CLINICAL TRIAL: NCT03764449
Title: A Single-Center, Non-Randomized, Open-Label, Parallel Group, Two-Treatment Study Investigating the Absolute Oral Bioavailability of Balovaptan After Single and Multiple Daily Oral Doses of Balovaptan in Healthy Volunteers
Brief Title: A Study Investigating the Absolute Oral Bioavailability of Balovaptan After Single and Multiple Daily Oral Doses of Balovaptan in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WP40607
Record Dates: First submitted 2018-11-30; First posted 2018-12-05 (Actual); Results first posted 2020-02-24 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — balovaptan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Participants received the study drug at dose level A in 2 periods. There was a minimum of a 14-day wash out period between Day 1 of Period 1 and Day 1 of Period 2.
  Interventions: Drug: Oral Balovaptan; Drug: IV Balovaptan
- Cohort 2 (Experimental): Participants received the study drug at dose level B in 2 periods. There was a minimum of a 14-day wash out period between Day 1 of Period 1 and Day 1 of Period 2.
  Interventions: Drug: Oral Balovaptan; Drug: IV Balovaptan

INTERVENTIONS:
Drug: Oral Balovaptan — In Period 1, balovaptan was administered as a single oral dose.
  In Period 2, balovaptan was administered as an oral dose once daily on Day 1 to Day 14.
Drug: IV Balovaptan — In Period 1, IV infusion of balovaptan was administered after the balovaptan oral dose.
  In Period 2, IV infusion of balovaptan was administered after the final oral dose of balovaptan.

SUMMARY:
This study was a non-randomized, open-label, parallel group, two-treatment study in healthy volunteers to investigate the absolute oral bioavailability of balovaptan. The study was conducted at 1 site in the Netherlands.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects. Healthy status is defined by absence of evidence of any active or chronic disease following a detailed medical and surgical history, a complete physical examination including vital signs, 12-lead ECG, hematology, blood chemistry, urinalysis, and serology.
* Body Mass Index of 18 to 30 kg/m2, inclusive.
* For women of childbearing potential: agreement to use at least 2 acceptable contraceptive methods during the treatment period and for 90 days after the last dose of study drug.
* For men: agreement to use contraceptive measures, and agreement to refrain from donating sperm until 90 days after the last dose of study drug.

Exclusion Criteria:

* Female subjects who are pregnant or lactating.
* Any condition or disease detected during the medical interview/physical examination that would render the subject unsuitable for the study, place the subject at undue risk or interfere with the ability of the subject to complete the study in the opinion of the Investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2019-03-04 (Actual); Study Completion 2019-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Pra International Group B.V, Groningen, Netherlands

REFERENCES:
- [Derived] Derks M, Lennon-Chrimes S, Guenther A, Squassante L, Wandel C, Szczesny P, Paehler A, Kletzl H. Bioavailability and pharmacokinetic profile of balovaptan, a selective, brain-penetrant vasopressin 1a receptor antagonist, in healthy volunteers. Expert Opin Investig Drugs. 2021 Aug;30(8):893-901. doi: 10.1080/13543784.2021.1948009. Epub 2021 Jul 16. PMID 34176392

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 1 site in the Netherlands.
Pre-assignment Details: Participants in this study included healthy volunteers.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.4 (16.18) | 33.5 (13.24) | 37.4 (14.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 6 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 8 | 6 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 8 | 14
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Absolute Bioavailability of Oral Balovaptan at Dose Level A (Cohort 1)
Description: Absolute oral bioavailability of a single dose A of balovaptan.
Time Frame: Day 1 of Period 1 (Period 1 is 14 days).
Population: The Pharmacokinetic (PK) analysis population consisted of all participants who received at least one dose of balovaptan. Participants were excluded from the PK analysis population if they significantly violated the inclusion or exclusion criteria, deviated significantly from the protocol, or if data were unavailable or incomplete.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage
Arm/Group | Cohort 1
Number analyzed (Participants) | 8
Percentage | 100.6 (31.4)

2. Secondary Outcome: Absolute Bioavailability of Oral Balovaptan at Dose Level B (Cohort 2)
Description: Absolute oral bioavailability of a single dose B balovaptan.
Time Frame: Day 1 of Period 1 (Period 1 is 14 days).
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage
Arm/Group | Cohort 2
Number analyzed (Participants) | 8
Percentage | 108.2 (5.9)

3. Secondary Outcome: Absolute Bioavailability of Oral Balovaptan at Dose A and Dose B
Description: Absolute oral bioavailability of balovaptan after once daily doses of Dose A and Dose B for 14 days.
Time Frame: Day 14 of Period 2 (Period 2 is 19 days).
Population: PK analysis consisted of all receiving at least 1 dose balovaptan.Participants excluded from analysis, if significantly violated inclusion/exclusion criteria, deviated significantly from protocol, or if data unavailable/incomplete.There were 2 outliers;sensitivity analysis excluding those 2,resulted in similar bioavailability across all treatments.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
Percentage | 82.3 (72.4) | 103.1 (4.1)

4. Secondary Outcome: Maximum Plasma Concentration (Cmax) of IV Balovaptan
Time Frame: Day 1 of Period 1 (Period 1 is 14 days); Day 14 of Period 2 (Period 2 is 19 days).
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
pg/mL
  Day 1 of Period 1 | 688 (30.5) | 1601 (28.2)
  Day 14 of Period 2 | 1591 (115.8) | 1974 (37.9)

5. Secondary Outcome: Cmax of Oral Balovaptan
Time Frame: Day 1 of Period 1 (Period 1 is 14 days); Day 14 of Period 2 (Period 2 is 19 days).
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
ng/mL
  Day 1 of Period 1 | 36.9 (36.8) | 443 (15.2)
  Day 14 of Period 2 | 108 (20.4) | 643 (25.0)

6. Secondary Outcome: Cmax of M2 Metabolites
Time Frame: Day 1 of Period 1 (Period 1 is 14 days); Day 14 of Period 2 (Period 2 is 19 days).
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
ng/mL
  Day 1 of Period 1 | 3.87 (62.1) | 23.6 (38.1)
  Day 14 of Period 2 | 20.3 (65.8) | 105 (29.0)

7. Secondary Outcome: Cmax of M3 Metabolites
Time Frame: Day 1 of Period 1 (Period 1 is 14 days); Day 14 of Period 2 (Period 2 is 19 days).
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
ng/mL
  Day 1 of Period 1 | 6.18 (28.6) | 57.9 (30.3)
  Day 14 of Period 2 | 57.2 (18.8) | 260 (26.5)

8. Secondary Outcome: Time to Maximum Observed Plasma Concentration (Tmax) of IV Balovaptan
Time Frame: Day 1 of Period 1 (Period 1 is 14 days); Day 14 of Period 2 (Period 2 is 19 days).
Population: The Pharmacokinetic (PK) analysis population consisted of all partcipants who received at least one dose of balovaptan. Participants were excluded from the PK analysis population if they significantly violated the inclusion or exclusion criteria, deviated significantly from the protocol, or if data were unavailable or incomplete.
Measure: Median (Full Range); unit: Hour
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
Hour
  Day 1 of Period 1 | 0.25 [0.10 to 0.25] | 0.25 [0.25 to 0.25]
  Day 14 of Period 2 | 0.25 [0.25 to 14.8] | 0.25 [0.25 to 1.00]

9. Secondary Outcome: Tmax of Oral Balovaptan
Time Frame: Day 1 of Period 1 (Period 1 is 14 days); Day 14 of Period 2 (Period 2 is 19 days).
Population: as for outcome 1
Measure: Median (Full Range); unit: Hour
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
Hour
  Day 1 of Period 1 | 1.23 [0.50 to 1.35] | 1.00 [1.00 to 1.33]
  Day 14 of Period 2 | 1.28 [0.50 to 1.75] | 1.11 [0.50 to 1.75]

10. Secondary Outcome: Tmax of M2 Metabolites
Time Frame: Day 1 of Period 1 (Period 1 is 14 days); Day 14 of Period 2 (Period 2 is 19 days).
Population: as for outcome 1
Measure: Median (Full Range); unit: Hour
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
Hour
  Day 1 of Period 1 | 24.0 [24.0 to 48.0] | 24.0 [16.0 to 24.1]
  Day 14 of Period 2 | 4.50 [1.22 to 12.0] | 3.38 [1.22 to 6.00]

11. Secondary Outcome: Tmax of M3 Metabolites
Time Frame: Day 1 of Period 1 (Period 1 is 14 days); Day 14 of Period 2 (Period 2 is 19 days).
Population: as for outcome 1
Measure: Median (Full Range); unit: Hour
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
Hour
  Day 1 of Period 1 | 48.0 [16.0 to 60.0] | 12.0 [4.50 to 24.1]
  Day 14 of Period 2 | 2.13 [1.00 to 4.50] | 1.88 [1.22 to 4.50]

12. Secondary Outcome: Apparent Terminal Half-Life (t1/2) of IV Balovaptan
Time Frame: Day 1 of Period 1 (Period 1 is 14 days); Day 14 of Period 2 (Period 2 is 19 days).
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
Hour
  Day 1 of Period 1 | 35.2 (23.7) | 19.5 (34.0)
  Day 14 of Period 2 | 27.7 (18.3) | 15.7 (28.2)

13. Secondary Outcome: T1/2 of Oral Balovaptan
Time Frame: Day 1 of Period 1 (Period 1 is 14 days); Day 14 of Period 2 (Period 2 is 19 days).
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
Hour
  Day 1 of Period 1 | 38.8 (25.9) | 29.1 (28.7)
  Day 14 of Period 2 | 31.2 (15.6) | 22.7 (15.7)

14. Secondary Outcome: T1/2 of M2 Metabolites
Time Frame: Day 1 of Period 1 (Period 1 is 14 days); Day 14 of Period 2 (Period 2 is 19 days).
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
Hour
  Day 1 of Period 1 | 48.5 (36.7) | 35.7 (27.2)
  Day 14 of Period 2 | 36.3 (25.0) | 28.5 (13.5)

15. Secondary Outcome: T1/2 of M3 Metabolites
Time Frame: Day 1 of Period 1 (Period 1 is 14 days); Day 14 of Period 2 (Period 2 is 19 days).
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
Hour
  Day 1 of Period 1 | 93.0 (18.5) | 68.2 (29.8)
  Day 14 of Period 2 | 60.3 (29.1) | 33.7 (11.2)

16. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to the Last Measurable Plasma Concentration Time Point (AUC0-last) of IV Balovaptan
Time Frame: Day 1 of Period 1 (Period 1 is 14 days)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
h*pg/mL | 8087 (35.5) | 9372 (19.3)

17. Secondary Outcome: AUC0-last of Oral Balovaptan
Time Frame: Day 1 of Period 1 (Period 1 is 14 days)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
h*ng/mL | 937 (25.6) | 5497 (23.9)

18. Secondary Outcome: AUC0-last of M2 Metabolites
Time Frame: Day 1 of Period 1 (Period 1 is 14 days)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
h*ng/mL | 297 (72.0) | 1751 (37.5)

19. Secondary Outcome: AUC0-last of M3 Metabolites
Time Frame: Day 1 of Period 1 (Period 1 is 14 days)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
h*ng/mL | 754 (24.3) | 3908 (24.5)

20. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of IV Balovaptan
Time Frame: Day 1 of Period 1 (Period 1 is 14 days); Day 14 of Period 2 (Period 2 is 19 days).
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
h*pg/mL
  Day 1 of Period 1 | 8929 (34.0) | 9569 (19.8)
  Day 14 of Period 2 | 15492 (71.5) | 10430 (27.9)

21. Secondary Outcome: AUC0-inf of Oral Balovaptan
Time Frame: Day 1 of Period 1 (Period 1 is 14 days).
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
h*ng/mL | 1008 (24.4) | 5550 (23.9)

22. Secondary Outcome: AUC0-inf of M2 Metabolites
Time Frame: Day 1 of Period 1 (Period 1 is 14 days).
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
h*ng/mL | 520 (55.1) | 1819 (36.5)

23. Secondary Outcome: AUC0-inf of M3 Metabolites
Time Frame: Day 1 of Period 1 (Period 1 is 14 days).
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
h*ng/mL | 1122 (14.8) | 4221 (27.5)

24. Secondary Outcome: Area Under the Plasma Concentration-Time Curve Over the Dosing Interval at Steady State (AUC0-24) of IV Balovaptan
Time Frame: Day 1 of Period 1 (Period 1 is 14 days); Day 14 of Period 2 (Period 2 is 19 days).
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
h*pg/mL
  Day 1 of Period 1 | 4400 (42.8) | 6690 (13.9)
  Day 14 of Period 2 | 9898 (89.0) | 7908 (19.4)

25. Secondary Outcome: AUC0-24 of Oral Balovaptan
Time Frame: Day 1 of Period 1 (Period 1 is 14 days); Day 14 of Period 2 (Period 2 is 19 days).
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
h*ng/mL
  Day 1 of Period 1 | 458 (22.3) | 3632 (15.6)
  Day 14 of Period 2 | 1322 (19.3) | 5505 (30.7)

26. Secondary Outcome: AUC0-24 of M2 Metabolites
Time Frame: Day 1 of Period 1 (Period 1 is 14 days); Day 14 of Period 2 (Period 2 is 19 days).
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
h*ng/mL
  Day 1 of Period 1 | 54.7 (73.5) | 427 (41.1)
  Day 14 of Period 2 | 404 (64.2) | 2087 (32.1)

27. Secondary Outcome: AUC0-24 of M3 Metabolites
Time Frame: Day 1 of Period 1 (Period 1 is 14 days); Day 14 of Period 2 (Period 2 is 19 days).
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
h*ng/mL
  Day 1 of Period 1 | 106 (40.5) | 1188 (29.2)
  Day 14 of Period 2 | 1102 (17.4) | 4727 (28.3)

28. Secondary Outcome: Last Measurable Plasma Concentration (Clast) of IV Balovaptan
Time Frame: Day 1 of Period 1 (Period 1 is 14 days); Day 14 of Period 2 (Period 2 is 19 days).
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
pg/mL
  Day 1 of Period 1 | 13.6 (49.7) | 6.62 (29.8)
  Day 14 of Period 2 | 12.5 (45.5) | 6.92 (22.6)

29. Secondary Outcome: Clast of Oral Balovaptan
Time Frame: Day 1 of Period 1 (Period 1 is 14 days); Day 14 of Period 2 (Period 2 is 19 days).
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
ng/mL
  Day 1 of Period 1 | 1.22 (13.4) | 1.22 (10.6)
  Day 14 of Period 2 | 3.51 (62.2) | 3.40 (88.6)

30. Secondary Outcome: Clast of M2 Metabolites
Time Frame: Day 1 of Period 1 (Period 1 is 14 days); Day 14 of Period 2 (Period 2 is 19 days).
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
ng/mL
  Day 1 of Period 1 | 1.24 (10.4) | 1.25 (15.6)
  Day 14 of Period 2 | 3.19 (51.2) | 9.95 (58.0)

31. Secondary Outcome: Clast of M3 Metabolites
Time Frame: Day 1 of Period 1 (Period 1 is 14 days); Day 14 of Period 2 (Period 2 is 19 days).
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
ng/mL
  Day 1 of Period 1 | 1.43 (24.4) | 2.74 (55.8)
  Day 14 of Period 2 | 11.9 (21.3) | 17.6 (64.0)

32. Secondary Outcome: Time of Last Measurable Plasma Concentration (Tlast) of IV Balovaptan
Time Frame: Day 1 of Period 1 (Period 1 is 14 days); Day 14 of Period 2 (Period 2 is 19 days).
Population: as for outcome 1
Measure: Median (Full Range); unit: Hour
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
Hour
  Day 1 of Period 1 | 106.75 [106.75 to 106.82] | 100.75 [58.75 to 106.75]
  Day 14 of Period 2 | 106.75 [106.75 to 106.77] | 82.75 [58.75 to 106.75]

33. Secondary Outcome: Tlast of Oral Balovaptan
Time Frame: Day 1 of Period 1 (Period 1 is 14 days); Day 14 of Period 2 (Period 2 is 19 days).
Population: as for outcome 1
Measure: Median (Full Range); unit: Hour
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
Hour
  Day 1 of Period 1 | 132.00 [108.00 to 168.05] | 156.00 [96.00 to 216.03]
  Day 14 of Period 2 | 108.00 [108.00 to 108.02] | 108.00 [108.00 to 108.02]

34. Secondary Outcome: Tlast of M2 Metabolites
Time Frame: Day 1 of Period 1 (Period 1 is 14 days); Day 14 of Period 2 (Period 2 is 19 days).
Population: as for outcome 1
Measure: Median (Full Range); unit: Hour
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
Hour
  Day 1 of Period 1 | 120.00 [72.00 to 168.32] | 168.00 [144.00 to 216.00]
  Day 14 of Period 1 | 108.00 [108.00 to 108.02] | 108.00 [108.00 to 108.02]

35. Secondary Outcome: Tlast of M3 Metabolites
Time Frame: Day 1 of Period 1 (Period 1 is 14 days); Day 14 of Period 2 (Period 2 is 19 days).
Population: as for outcome 1
Measure: Median (Full Range); unit: Hour
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
Hour
  Day 1 of Period 1 | 216.00 [192.00 to 216.05] | 216.00 [192.00 to 216.03]
  Day 14 of Period 2 | 108.00 [108.00 to 108.02] | 108.00 [108.00 to 108.02]

36. Secondary Outcome: Terminal Elimination Rate Constant (λz) of IV Balovaptan
Time Frame: Day 1 of Period 1 (Period 1 is 14 days); Day 14 of Period 2 (Period 2 is 19 days).
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: /hour
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
/hour
  Day 1 of Period 1 | 0.0197 (23.7) | 0.0356 (34.0)
  Day 14 of Period 2 | 0.0250 (18.3) | 0.0442 (28.2)

37. Secondary Outcome: λz of Oral Balovaptan
Time Frame: Day 1 of Period 1 (Period 1 is 14 days); Day 14 of Period 2 (Period 2 is 19 days).
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: /h
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
/h
  Day 1 of Period 1 | 0.0179 (25.9) | 0.0239 (28.7)
  Day 14 of Period 2 | 0.0222 (15.6) | 0.0306 (15.7)

38. Secondary Outcome: λz of M2 Metabolites
Time Frame: Day 1 of Period 1 (Period 1 is 14 days); Day 14 of Period 2 (Period 2 is 19 days).
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: /hour
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
/hour
  Day 1 of Period 1 | 0.0143 (36.7) | 0.0194 (27.2)
  Day 14 of Period 2 | 0.0191 (25.0) | 0.0244 (13.5)

39. Secondary Outcome: λz of M3 Metabolites
Time Frame: Day 1 of Period 1 (Period 1 is 14 days); Day 14 of Period 2 (Period 2 is 19 days).
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: /hour
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
/hour
  Day 1 of Period 1 | 0.0075 (18.5) | 0.0102 (29.8)
  Day 14 of Period 2 | 0.0115 (29.1) | 0.0206 (11.2)

40. Secondary Outcome: Total Body Clearance (CL) of IV Balovaptan
Time Frame: Day 1 of Period 1 (Period 1 is 14 days); Day 14 of Period 2 (Period 2 is 19 days).
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
L/h
  Day 1 of Period 1 | 9.98 (34.1) | 9.75 (20.4)
  Day 14 of Period 2 | 6.23 (71.4) | 9.36 (27.1)

41. Secondary Outcome: Volume of Distribution (Vss) of IV Balovaptan
Time Frame: Day 1 of Period 1 (Period 1 is 14 days); Day 14 of Period 2 (Period 2 is 19 days).
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
Liter
  Day 1 of Period 1 | 396 (53.1) | 197 (21.9)
  Day 14 of Period 2 | 166 (95.4) | 154 (15.3)

42. Secondary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events
Time Frame: Up to 35 days from screening (sceening is up to 28 days prior to admission to the clinical research unit).
Population: The safety analysis population consisted of participants who received at least one dose of balovaptan.
Measure: Number; unit: Percentage
Groups:
- Cohort 1, Period 1; Cohort 1, Period 2: Participants received the study drug at dose level A in 2 periods. There was a minimum of a 14-day wash out period between Day 1 of Period 1 and Day 1 of Period 2.
- Cohort 2, Period 1; Cohort 2, Period 2: Participants received the study drug at dose level B in 2 periods. There was a minimum of a 14-day wash out period between Day 1 of Period 1 and Day 1 of Period 2.
Arm/Group | Cohort 1, Period 1 | Cohort 1, Period 2 | Cohort 2, Period 1 | Cohort 2, Period 2
Number analyzed (Participants) | 8 | 8 | 8 | 8
Percentage | 50 | 75 | 63 | 88

ADVERSE EVENTS:
Time Frame: Up to 21 days postdose (15 March 2019).
Groups:
- Cohort 1 Period 1: Balovaptan was administered at dose level A as a single oral dose. IV infusion of balovaptan was administered after the balovaptan oral dose.
- Cohort 1, Period 2: Balovaptan was administered at dose level A as an oral dose once daily on Day 1 to Day 14. IV infusion of balovaptan was administered after the final oral dose of balovaptan.
- Cohort 2, Period 1: Balovaptan was administered as a single oral dose at dose level B. IV infusion of balovaptan was administered after the balovaptan oral dose.
- Cohort 2, Period 2: Balovaptan was administered at Dose level B as an oral dose once daily on Day 1 to Day 14. IV infusion of balovaptan was administered after the final oral dose of balovaptan.
Arm/Group | Cohort 1 Period 1 | Cohort 1, Period 2 | Cohort 2, Period 1 | Cohort 2, Period 2
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 4/8 | 6/8 | 5/8 | 7/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 Period 1 (N=8) | Cohort 1, Period 2 (N=8) | Cohort 2, Period 1 (N=8) | Cohort 2, Period 2 (N=8)
Ear congestion (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site haematoma (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Catheter site swelling (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Infusion site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (3)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Mood altered (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nightmare (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-10-22): https://cdn.clinicaltrials.gov/large-docs/49/NCT03764449/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-27): https://cdn.clinicaltrials.gov/large-docs/49/NCT03764449/SAP_001.pdf